CLINICAL TRIAL: NCT07214051
Title: PR-CEAL: Community Outreach Engagement Group
Acronym: PR-CEAL:COEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Vivian Colon Lopez, Principal Investigator, University of Puerto Rico Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2410002304; SUB-OTA No. 6922-03-COVID-S026 (Other Grant/Funding Number: WESTAT, INC)
Record Dates: First submitted 2025-09-19; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Prevention; Colorectal Cancer Prevention; Cervical Cancer Prevention
Keywords: Breast Cancer Screening Test; Colorectal Cancer Screening Test; Cervical Cancer Screening Test; Puerto Rico; overdue cancer screening

STUDY DESIGN:
Intervention Model Description: This study recruited 500 participants, allocated on 1:1 ratio for intervention or control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity and Mental Health Information (No Intervention): The control group (n=250) received physical activity and mindfulness materials. Two follow-up calls, at four- week intervals each, assessed screening status for all participants. Once the study concluded, cancer information was sent to participants by certified mail.
- Cancer Screening Information (Experimental): The intervention group (n=250) received educational materials that included: screening center details, and reminders related to cancer screening. Two follow-up calls, at four-week intervals each, assessed screening status for all participants.
  Interventions: Behavioral: Cancer Screening Information

INTERVENTIONS:
Behavioral: Cancer Screening Information — The intervention group (n=250) received educational materials that included: screening center details, and reminders related to cancer screening. Two follow-up calls, at four-week intervals each, assessed screening status for all participants.
  Arms: Cancer Screening Information

SUMMARY:
The United States Preventive Services Task Force (USPSTF) recommends regular screenings for breast, cervical, and colorectal cancer. The COVID-19 pandemic has disrupted health screening practices, leading to a decrease in cancer screenings among the United States including Puerto Rico. This has been attributed to unwillingness, distrust, and insecurity related to accessing healthcare services. To overcome these challenges, a collaboration between PR-CEAL's Community Outreach Engagement Group (COEG), academic researchers, healthcare institutions, and community-based organizations proposed to engage in different community activities throughout the island. In these events, investigators conducted a single blinded community-based Randomized Clinical Trial (RCT) regarding cancer screening practices in women 21 through 75 years. The community-based RCT employed a mixed-method design to gain insights into the perception of health and cancer screening status of participants regarding breast, uterine (cervical), and colorectal cancer. Data was collected through in person interviews and two follow up phone calls, enabling the researchers to obtain valuable sociodemographic information, assessing cancer screening history, and identifying existing barriers.

The hypothesis of this study is that implementing evidence-based intervention at community settings across Puerto Rico will have a significant positive effect on cancer screening rates among non-adherent patients. By identifying and adapting the Prevention Care Management for Cancer Screening intervention and leveraging the expertise of the National Cancer Institute, the study aimed to improve screening rates, address barriers that hinder or delay screenings, and raise awareness about the importance of early detection.

DETAILED DESCRIPTION:
The study aimed to recruit 500 participants. Recruited participants were women aged 21 through 75 years, overdue in at least one cancer screening test (breast cancer, cervical cancer, and/or colorectal cancer) based on the US Preventive Services Task Force (USPSTF) guidelines. Once the woman verbally consents to participate in the RCT, four pre-screening questions and a Cancer Screening Module will be conducted to determine her eligibility. If the woman is eligible, informed consent will be completed, followed by a contact information module, and a baseline survey using an adaptation of the Prevention Care Management approach.

After identifying overdue participants and obtaining their RCT participation consent, REDcap randomly assigned them to control or intervention groups in a 1:1 ratio. The control group (n=250) received physical activity and mindfulness materials, while the intervention group (n=250) received educational materials that included screening center details and reminders related to cancer screening. Two follow-up calls, at four-week intervals, were performed to assess the screening status for all participants.

1. If the initial call was unanswered, two more attempts were made on consecutive days. Voicemails, if possible, will prompt a response. A second follow-up call was made four weeks later to evaluate the status.
2. If a participant answers the initial call but remains unscreened, Health Promoter encourages the intervention group to schedule doctor visits and cancer screening appointments. The second follow-up call in four weeks assesses the status. If the initial call is unanswered, two more attempts follow. Voicemails may be used to prompt a response.
3. If the participant answered the initial call and has an appointment for cancer screening, a second follow-up call in four weeks will assess screening status. If the initial call was unanswered, two more attempts were made. Voicemails were used to prompt a response.
4. The intervention ended if the participant confirmed an up-to-date status in the initial call.

Once the study concluded, the control group received the cancer educational materials by mail.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Between 21 and 75 years old
* Participant is overdue in at least one cancer screening (breast, cervical or colorectal), according to the USPTF guidelines.
* Participants that have not reported any cognitive, mental or physical limitation.
* Ability to read.
* Access to a telephone.
* Participants that are not in active cancer treatment.

Exclusion Criteria:

* Male
* Women younger than 21 years or older than 75 years.
* Participants that are not overdue in any cancer screening (breast, cervical or colorectal), according to the USPTF guidelines.
* Participants that are cognitive, mental or physically limited.
* Participants who are not able to read.
* Participants who don't have access to a telephone.
* Participants that are in active cancer treatment.

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who compelled with cancer screening test | Eight weeks
  Once recruited, participants have two follow-up calls at four-week intervals each to assess their cancer screening test status (i.e., whether they have had their mammograms, pap test, and FOBT or colonoscopy).

SECONDARY OUTCOMES:
Number of participants that scheduled an appointment for cancer screening | Eight weeks
  Once recruited, participants have two follow-up calls at four-week intervals each to assess the scheduling of an appointment for their cancer screening test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico, Comprehensive Cancer Center, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided